CLINICAL TRIAL: NCT03268759
Title: Development of Reward Processing in Prenatally Exposed Adolescents and Young Adults
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0203014534; 1K01DA042937 (NIH)
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Pre-natal Cocaine Exposure; Risk-Taking
Keywords: substance abuse
MeSH Terms: conditions — Risk-Taking; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCE: Emerging adult individuals who were exposed to cocaine in-utero
  Interventions: Other: fMRI
- NCE: Emerging adult individuals who were not exposed to cocaine in-utero
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — Observation of neural markers of reward processing
  Other Names: EEG

SUMMARY:
Reward processing will be examined in prenatally exposed emerging adults in a longitudinal design. Participants will be followed for one year to see if neural markers of reward processing prospectively predict risk-taking behavior.

DETAILED DESCRIPTION:
This cohort will be drawn from a pre-existing cohort of individuals recruited as part of an already existing study, and who have been followed since birth. Reward processing will be measured in two temporally close testing sessions involving two methodologies, electrophysiology and fMRI. Information will also be collected pertaining to experimental and problematic drug use, as well as information about mood, at the recording sessions. Drug use and mood information will then be collected once again in quarterly follow-up sessions for one year. The goal is to examine if PCE status and reward processing are risk factors for problematic drug abuse and risky behaviors in emerging adulthood, and if these factors interact to increase such risk.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and to comply with all study procedures.
2. Healthy emerging adults between 18-20 years of age (the age of the currently followed sample at the time of the proposed start date).

Exclusion Criteria:

* 1. A serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain. 2. A medical condition that requires treatment with a medication with psychotropic effects.

  3. Evidence of stroke or space occupying lesions observed on conventional, clinical MR images.

  4. Any contraindications to MRI scanning (i.e., metal implants, pacemakers, etc.) 5. History of loss of consciousness (LOC) for longer than 30 minutes or LOC with any neurological sequelae.

  6. DSM-5 criteria for intellectual disability. 7. Current or a history of active neurological or psychiatric disorders, such as psychosis, bipolar illness, major depression, organic brain disease, dementia or DSM-V Axis I Psychiatric Disorder, including current alcohol or substance disorders. Participants will not be excluded for substance or alcohol use, only the presence of substance disorders.

  8. Current pregnancy. Female participants will be excluded if they report being currently pregnant or present positive for pregnancy after being given a urine test at the time of recruitment or scanning. If they become pregnant during the one-year follow-up duration of the study after the MRI scan is completed, they will remain in the study for the quarterly follow-ups and be referred to pre-natal care if they have not begun such care already.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Emerging adults in this study will be drawn from a sample of 359 individuals who have been participating in a longitudinal study of the effects of PCE on physical, social, cognitive and emotional development. Children and their mothers who were exposed to drugs other than cocaine were also enrolled, as were non-drug exposed controls. Prenatal drug exposure status was ascertained at time of recruitment via a detailed interview that covered lifetime substance use and use in the past 30 days, as well as a urine screening of mother and infant and meconium toxicology. The sample from which participants will be recruited consists of 81% African American, 6.5% Hispanic and 12.5% Caucasian children, all of who come from the greater New Haven area. The sample was recruited at birth over a 5-year period.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Change in Risk-taking behavior:Drug and alcohol use | 4x per year for one year (Baseline, 4 months, 8 months, 12 months)
  Teen Addiction Severity Index (Interview)
Change in Risk-taking behavior:gambling behaviors | 4x per year for one year (Baseline, 4 months, 8 months, 12 months)
  Massachusetts gambling screen (MAGS)

SECONDARY OUTCOMES:
Change in affect over time | 4x per year for one year (Baseline, 4 months, 8 months, 12 months)
  Positive and Negative Affect Scales (PANAS)
Change in alexithymia over time | 4x per year for one year (Baseline, 4 months, 8 months, 12 months)
  Toronto Alexithymia Scale (TAS-20)
Change in experience of reward | 4x per year for one year (Baseline, 4 months, 8 months, 12 months)
  Chapman Social and Physical Anhedonia Questionnaires
Change in emotion regulation strategies | 4x per year for one year (Baseline, 4 months, 8 months, 12 months)
  Emotion regulation questionaire (ERQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No